CLINICAL TRIAL: NCT03721471
Title: Outcome of Very Old Patients Admitted for Elective Major Surgery, the Effect of Frailty
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/315
Record Dates: First submitted 2018-10-02; First posted 2018-10-26 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2022-11

CONDITIONS: Frail Elderly Syndrome; Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Frail, non-frail: Frail Group: Those individuals identified as frail by low hand-grip-strength and/or the Clinical Frailty Scale.
  Non-frail Group: Those individuals identified as not frail by hand-grip-strength and/or the Clinical Frailty Scale.
  Interventions: Other: Scoring of frailty

INTERVENTIONS:
Other: Scoring of frailty — 1. Patients will be scored by the Clinical frailty Scale
  2. Patients' hand-grip-strength will be measured by a dynamometer.

SUMMARY:
The aim of the study is to investigate the effect of frailty in patients ≥ 80 years admitted for elective major abdominal surgery.

DETAILED DESCRIPTION:
Patients ≥ 80 years admitted for elective major abdominal surgery will be asked to participate in this study where frailty will be scored using the Clinical Frailty Scale and by measuring hand-grip-strength.

Primary outcome is mortality at 30 days, 90 days and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* age 80 years or above
* elective abdominal surgery
* informed consent

Exclusion Criteria:

* age less than 80 years
* emergency surgery
* palliative surgery ( e.g performing entero-enteroanastomosis to relieve obstruction)

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 80 years admitted for elective major abdominal surgery at Haukeland University Hospital, Bergen, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Time to death | Up to one year
  Time until subject dies or up to one year after surgery

SECONDARY OUTCOMES:
Postoperative complications | Up to 90 days after surgery
  Complications as graded by the Clavien-Dindo system and defined by the EPCO-definitions.
Discharge to institution | Up to 90 days after surgery
  Discharge to nursing home
Worsening functional status | 1 year postoperatively.
  Increased need of assistance in performing ADL.
Mortality at 30 days | 30 days after surgery
  Death within 30 days after surgery
Mortality at 90 days | 90 days after surgery
  Death within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ib Jammer, PhD, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers